CLINICAL TRIAL: NCT01662557
Title: Treatment of Early Childhood Overweight in Primary Care: Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Geisinger Center for Health Research (Unknown); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 807610; R34DK080473 (NIH)
Record Dates: First submitted 2012-08-07; First posted 2012-08-10 (Estimated); Last update posted 2012-08-15 (Estimated); Status verified 2011-01

CONDITIONS: Obesity
Keywords: Pediatric Obesity
MeSH Terms: conditions — Obesity; Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Family Behavior Modification (Active Comparator): Family-based behavior modification with parent and child using goal setting, self monitoring, reinforcement, behavioral skills training, and tasting opportunities.
  Interventions: Behavioral: Family Behavior Modification
- Minimal Nutrition Information (Other): Weekly mailings emphasizing healthy eating guidelines for families.
  Interventions: Other: Minimal Nutrition Information

INTERVENTIONS:
Behavioral: Family Behavior Modification — 5-month intervention for parents and children providing 15 sessions in behavioral skills training in self monitoring, Traffic Light Diet, goal setting, reinforcement and tasting sessions. Of the 15 sessions, 3 were structured as phone sessions.
  Other Names: FBM
  Arms: Family Behavior Modification
Other: Minimal Nutrition Information — Families assigned to MNI received a series of 15 mailings on topics related identifying a healthy body weight for children; energy balance and calorie requirements for children; MyPyramid for Kids; portion control; the benefits of physical activity and screen-time reduction; encouraging fruit and vegetable consumption; healthy snacks and smart shopping; and encouraging family meals.
  Other Names: MNI
  Arms: Minimal Nutrition Information

SUMMARY:
Childhood overweight continues to increase at an alarming rate and the need exists to find effective, accessible intervention strategies to prevent and treat children who are at risk for being overweight or are already overweight. The primary care setting provides an attractive option for families wishing to receive treatment, yet little is known about the feasibility, acceptance or efficacy of this intervention setting. The purpose of this study was to test two different primary care treatments that were intended to increase fruit and vegetable intake, increase physical activity, and reduce sedentary activity in children ages 4-8, who are overweight or at risk for becoming overweight. Both treatments involved the child and a parent/caregiver and both were conducted over a four month period. The parent/child dyads were selected from the pool of families who receive their primary care within the Geisinger Medical Center geographic area and who have been identified by their pediatrician as being overweight or at risk for becoming overweight (BMI >85th percentile for age). One group received weekly mailings which focused on healthy eating, promotion of fruit and vegetable intake and physical activity, and methods to reduce TV viewing time. The second group received a group-based intervention at one of the Geisinger Pediatric Clinic sites using specific behavioral strategies for increasing fruit and vegetable intake, reducing TV viewing and encouraging physical activity. Changes in overweight percentage, child BMI, lipid profile, glucose/insulin levels, and anthropometric measurements were analyzed, as well as treatment satisfaction and acceptance. The investigators hypothesized that children who receive Family Behavior Modification (FBM) in the primary care setting will show greater reductions in Body Mass Index (BMI), BMI z-score, percent overweight and waist circumference, and that children receiving FBM will show greater improvements in dietary intake, increased physical activity, reduced sedentary activity, and improvements in cardiovascular outcomes.

ELIGIBILITY:
Inclusion Criteria:

* 4-8 year old children
* overweight or obese (BMI≥85th percentile, based on age and sex)
* Parent/primary caregiver willing to attend sessions with child

Exclusion Criteria:

* Failure to meet BMI criteria
* Child with elevated internalizing or externalizing behavioral problems, as assessed through Child Behavior Checklist (CBCL)
* Elevated parent distress, as measured by Symptom Checklist-90 (SCL-90)
* Child on medications with any weight-altering effect
* Inability to participate in moderate physical activity or attend study visits
* Residing >1 hour from study site

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 51 (Actual)
Dates: Start 2008-02; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Child's Overweight Percentage | Baseline and Month 5
  Change in child's overweight percentage will be measured from baseline to end of treatment (month 5)
Body Mass Index z-score (BMI-z) | Baseline and Month 5
  Change in BMI-z score will be measured from baseline to end of treatment (month 5)
Waist Circumference | Baseline and Month 5
  Change in child's waist circumference will be measured from baseline to end of treatment (month 5).
Body Mass Index (BMI) | Baseline and Month 5
  Change in BMI will be measured from baseline to end of treatment (month 5).

SECONDARY OUTCOMES:
Dietary Intake | Baseline and Month 5
  Change in dietary intake (kcals, protein, fat, saturated fat, cholesterol, fiber, carbohydrate, fruit/veg servings, Vitamins A and C) will be assessed from baseline to end of treatment (month 5) using 24-hour recall interviews.
Activity Level | Baseline to Month 5
  Physical activity (sedentary, light, moderate and moderate to vigorous) will be assessed via accelerometry between baseline and end of treatment (month 5).
Insulin (uUnits/ml) | Baseline and Month 5
  Change in fasting insulin will be measured at baseline and end of treatment (month 5).
Glucose (mg/dl) | Baseline and Month 5
  Change in fasting glucose levels will be measured from baseline to end of treatment (month 5).
Triglycerides (mg/dl) | Baseline and Month 5
  Change in fasting triglyceride levels will be measured from baseline to end of treatment (month 5).
HDL (mg/dl) | Baseline and Month 5
  Change in HDL levels will be measured from baseline to end of treatment (month 5).
LDL (mg/dl) | Baseline and Month 5
  Change in LDL levels will be measured from baseline to end of treatment (month 5).

CONTACTS AND LOCATIONS:
Overall Officials: Myles S Faith, Ph.D., Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania Center for Weight and Eating Disorders, Philadelphia, Pennsylvania, United States